CLINICAL TRIAL: NCT06329206
Title: A Phase Ia/Ib Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Antitumor Activity of GH2616 Tablet in Subjects With Advanced Solid Tumors
Brief Title: A Phase Ia/Ib Study of GH2616 Tablet in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Hubei Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH2616-101
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GH2616 GROUP (Experimental): Dose Escalation: Dose Escalation Cohorts Subjects will be enrolled at various doses of GH2616. These Dose Escalation Cohorts will be utilized to To determine the maximum tolerated dose (MTD) and/or recommended dose for expansion(s) (RDEs) for Dose Expansion. Dose Escalation: Backfill Cohorts 2 ~ 3 dose cohorts are allowed to be backfilled.These Backfill Cohorts will be utilized to build additional data to support selection of doses and/or tumor types for further study in Dose Expansion.
  Dose Expansion: Expansion Cohorts 2 ~ 3 dose cohorts are planned.Subjects with advanced solid tumors harboring TP53 mutation and whole genome duplication (WGD+) will be enrolled.These Cohorts will be utilized to to determine the recommended Phase II dose (RP2D) of GH2616 Tablet.
  Interventions: Drug: GH2616 Tablets

INTERVENTIONS:
Drug: GH2616 Tablets — GH2616 tablets will be given orally

SUMMARY:
This is a Phase Ia/Ib, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, pharmacodynamics (PD) and preliminary efficacy of GH2616 Tablet in subjects with advanced solid tumors. It includes two parts: the dose escalation study (Phase Ia) and the dose expansion study (Phase Ib).

DETAILED DESCRIPTION:
Phase Ia: Dose Escalation Study This is a Phase Ia, open-label, multi-center, dose escalation study, aiming to investigate the safety, tolerability, PK, PD and preliminary anti-tumor activity of GH2616 Tablet in subjects with advanced solid tumors.

• Dose Escalation Phase This study will consist of 8, sequential, ascending-dose cohorts (A1~ A8) and utilize a "3+3" dose escalation design.

Phase Ib: Dose Expansion Study The Phase Ib part is an open-label, multi-center, dose expansion study, aiming to further evaluate the safety, tolerability, PK, PD, and preliminary anti-tumor activity of GH2616 Tablet in subjects with advanced solid tumors harboring TP53 mutation and WGD+ at the RDEs.

Phase Ib study will consist of 2 to 3 dose level cohorts (B1 ~ B3) of RDEs identified by the safety, tolerability, PK/PD characteristics, and preliminary efficacy data obtained from Phase Ia study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Men or women ≥18 years old.
  2. The following two points are evaluated by the Investigator and are deemed suitable to participate in the study: a. The subject fully understands the requirements of the study and voluntarily signs the written informed consent; b. Be able to comply with the medication requirements of the study and all study related procedures and evaluations.
  3. Meeting the requirements of tumor types shown below:

     Phase Ia Study:

     Subjects with a histological or cytological diagnosis of recurrent or metastatic advanced solid tumors who have failed or are intolerant to standard treatment, or have no standard therapy. The specific tumor types include but not limited to high-grade serous ovarian cancer (HGSOC), uterine carcinosarcoma (UCS), lung adenocarcinoma (LUAD), lung squamous cell carcinoma (LUSC), triple-negative breast cancer (TNBC), bladder urothelial carcinoma (BLCA), colorectal cancer (CRC), etc.

     Phase Ib study:

     Dose expansion study (Phase Ib): Subjects with a histological or cytological diagnosis of recurrent or metastatic advanced solid tumors harboring TP53 mutation and WGD+ who have failed or are intolerant to standard treatment, or have no standard therapy.

     The specific tumor types include but not limited to high-grade serous ovarian cancer (HGSOC), uterine carcinosarcoma (UCS), lung adenocarcinoma (LUAD), lung squamous cell carcinoma (LUSC), triple-negative breast cancer (TNBC), bladder urothelial carcinoma (BLCA), colorectal cancer (CRC), etc.. Note: The specific tumor types/basket design with specific gene(s) will be determined by the principal Investigator and the Sponsor based on the Phase Ia study results.
  4. Survival expectations are ≥ 12 weeks.
  5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 (Appendix 1).
  6. Subjects with advanced solid tumors have at least one evaluable lesion according to RECIST 1.1 (Appendix 2).
  7. Subjects with adequate organ function at the time of screening (requiring no blood transfusion, no use of hematopoietic stimulating factor or human albumin within 14 days prior to screening), specifically defined as:

     1. Blood routine: Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count (PLT) ≥100×109/L; Hemoglobin (HGB) ≥ 90 g/L (9 g/dL);
     2. Liver function: Serum Total bilirubin (TBIL) ≤ 1.5 Upper limit of normal value (ULN), and serum TBIL≤ 3×ULN in patients with liver metastasis or confirmed Gilbert syndrome. Alanine aminotransferase (ALT) and Aspartate transferase (AST) ≤ 2.5×ULN in subjects without liver metastasis; ALT or AST≤ 5×ULN in subjects with liver metastasis;
     3. Renal function: estimated creatinine clearance (CLcr) ≥ 60 mL/min as calculated using Cockcroft-Gault formula (Appendix 3);
     4. Coagulation function: Activated Partial thromboplastin Time (APTT) and international normalized ratio (INR) ≤ 1.5×ULN (or within target range if on anticoagulation therapy);
     5. Cardiac function: Echocardiography (ECHO) shows left ventricular ejection fraction (LVEF) > 50%.
  8. Serum pregnancy test (for female of childbearing potential) negative within 7 days prior to first dosing of study treatment. Male and female subjects of childbearing potential must agree to use effective methods of contraception throughout the study and for 3 months (male) or 6 months (female) after the last dose of the investigational product. A subject is of childbearing potential if, in the opinion of the Investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

* In Phase Ia and Ib studies, subjects will be excluded if they meet any of the following criteria:

  1. Has received chemotherapy within 21 days prior to the first administration of GH2616 Tablet or has received radiation therapy, biologic therapy, endocrine therapy, targeted therapy, immunotherapy, or other anti-tumor drug treatments within 28 days prior to the first administration of GH2616 Tablet, or other anti-tumor drugs or treatments within the following interval before the first administration of GH2616 Tablet: Nitrosoureas or mitomycin C within 6 weeks prior to the first administration of the investigational drug. Oral fluoropyrimidines, small molecule targeted therapies, and Chinese herbal medicines with indications for anti-tumor within 14 days prior to the first administration of the investigational drug. Local palliative radiation therapy within 14 days prior to the first administration of the investigational drug.
  2. Has received other investigational drugs or treatments not yet approved for marketing within 28 days prior to the first administration.
  3. Acute toxic effects of prior anti-tumor therapy have not recovered to clinically significant NCI-CTCAE V5.0 grade ≤ 1 toxicity or baseline specified in the inclusion criteria within 28 days prior to the first administration of GH2616 Tablet (excluding toxicities such as alopecia and fatigue that the Investigator deems to have no safety risk).
  4. At rest, the average Corrected QT interval (QTc, Fridericia's correction formula used) obtained by 12-lead Electrocardiograph (ECG) examination is > 450 ms for males or 470 ms for females (confirmed by repeated examinations). A variety of clinically significant arrhythmia, conduction, and resting ECG abnormalities, such as complete left bundle branch block, degree III, degree II, PR interval >250 ms. Various factors that may increase the risk of prolonged QTc or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome in a direct family member or sudden unexplained death before age 40, and use of any medications known to prolong QT intervals.
  5. Has evidence of infectious diseases:

     1. Active hepatitis B (hepatitis B surface antigen (HbsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV-DNA) > 500 IU/ml or 1000 cps/ml or lower limit of detection at the study site [only if lower limit of detection at the study site is higher than 500 IU/ml or 1000 cps/ml]), antiviral therapy other than interferon is allowed; active hepatitis C (subjects with hepatitis C virus (HCV) antibody positive but hepatitis C virus ribonucleic acid (HCVRNA) < lower limit of detection at the study site are allowed to be enrolled);
     2. HIV infected patients (HIV 1/2 antibody positive detected by antigen/antibody test); Considering that HIV infections can be chronically managed, expanding cancer clinical trial eligibility to be more inclusive of patients with HIV infections is justified in many cases, and may accelerate the development of effective therapies in cancer patients with these chronic infections. Therefore, well-controlled HIV patients who have been on established antiretroviral therapy (ART) for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment should be included. Note: patients who are using ART drugs that are prohibited or cautious concomitant medications specified in the protocol (e.g. strong inhibitors or strong inducers of P-gp) could be switched to an alternate effective ART regimen (with minimal drug-drug interaction potential) before study participation or should be excluded from the study if their regimen cannot be altered.
     3. Known active syphilis infection.
  6. Has symptomatic or active central nervous system (CNS) metastases. Treated or untreated asymptomatic patients with CNS lesions are eligible only if all of the following criteria are met:

     1. Presence of measurable lesions outside the CNS as determined by RECIST 1.1.
     2. No history of intracranial or spinal hemorrhage.
     3. No stereotactic radiation therapy or whole brain radiation therapy or neurosurgical resection within 28 days prior to initiation of study treatment.
     4. No continuous use of corticosteroids during CNS disease treatment period.
     5. Metastases limited to the cerebellum or supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
     6. No evidence of intermediate progression between completion of CNSdirected therapy (if given) and initiation of study treatment.
  7. Concurrent diseases that have not been controlled, such as:

     1. Severe infection, including but not limited to hospitalization due to infection, bacteremia, or severe pneumonia complications, occurs within 28 days prior to initiation of study treatment; Or patients who received therapeutic oral or intravenous antibiotics within 14 days prior to starting study treatment; Subjects receiving prophylactic antibiotics for needle biopsy can be included.
     2. Heart failure consistent with New York Heart Association Grades ≥ II within 6 months prior to initiation of study treatment.
     3. Other malignancies (other than in situ cancers such as non-melanoma basal cell carcinoma or squamous cell carcinoma of the skin, breast/cervical carcinoma in situ, superficial bladder carcinoma that have received radical treatment and no evidence of disease recurrence, etc.) within 5 years prior to initiation of treatment.
     4. Current subjects with cancerous meningitis, spinal cord compression, etc..
     5. Has a history of poorly controlled hypertension within 28 days prior to initiation of study treatment, defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, despite treatment with multiple antihypertensive medications.
     6. Any arterial thromboembolic event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, occurred within 6 months prior to initiation of study treatment.
     7. Significant malnutrition, such as the need for intravenous nutrient supplementation. Those who were stable for more than 28 days after correction of malnutrition before treatment of first dose of investigational product could be included.
     8. Tumor invasion of surrounding important organs or blood vessels (such as mediastinal great vessels, superior vena cava, trachea, esophagus, etc.), or at risk of esophagotracheal fistula or esophagopleural fistula.
     9. After endoesophageal or tracheal stent implantation.
     10. Has a history of gastrointestinal perforation and/or fistula 6 months prior to initiation of study treatment.
     11. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (monthly or more frequent).
     12. Uncontrolled tumor-related pain, or no stable pain regimen.
  8. Allergic to GH2616 Tablet or its components.
  9. Significant impairment of oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction, etc..
  10. Has severe lung disease or history, such as moderate to severe chronic obstructive pulmonary disease (COPD), evidence of interstitial lung disease (ILD)/pneumonitis on baseline imaging, history of ILD, drug-induced ILD, acute or chronic infectious pneumonia, lung transplantation, etc..
  11. Use of strong inhibitors or inducers of P-glycoprotein (P-gp) within 14 days or 5 halflives (whichever is longer) before the first administration (refer to Appendix 5).
  12. Use of sensitive narrow therapeutic index CYP3A4 substrate within 14 days or 5 halflives (whichever is longer) before the first administration (refer to Appendix 4).
  13. Pregnant or lactating women.
  14. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
  15. Has a major surgical procedure (craniotomy, thoracotomy, laparotomy, vascular intervention) within 28 days prior to the first administration, or had an unhealed wound, ulcer, or fracture. Note: For palliative care purposes, local surgical treatment of isolated lesions is acceptable.
  16. Has a clear history of mental disorder with ongoing treatment.
  17. Has a treatment history of KIF18A inhibitor.
  18. Subjects with POLE gene hotspot mutated, or hypermutator phenotype.
  19. In the opinion of the Investigator, there are other factors that the subject is unsuitable for participation in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Adverse Events (AEs) or Serious Adverse Events (SAEs) | 2 years
  Adverse events (AE), serious adverse events (SAE), and severity of AE using the NCI-CTCAE version 5.0.
Dose-limiting Toxicities Incidence Count Among Study Participant | 2 years
  DLT refers to Dose-Limiting Toxicity. It is defined as a side effect or adverse reaction of a drug or treatment that is severe enough to prevent an increase in dosage. Identifying DLT is crucial in clinical trials for determining the maximum tolerated dose (MTD) of a new drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) based on RECIST 1.1 criteria | 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR). (phase I)
Progression-Free Survival (PFS) based on RECIST 1.1 criteria | 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first. (phase I)
Duration of Response (DOR) based on RECIST 1.1 criteria | 2 years
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD). (phase I)
Plasma Concentration (Cmax) | 2 years
  Highest observed plasma concentration of GH2616. (phase I)
Area Under the plasma Concentration-Time Curve (AUC) | 2 years
  Area under the plasma concentration time curve of GH2616. (phase I)
Time to CAchieve Cmax (Tmax) | 2 years
  Time of highest observed plasma concentration of GH2616. (phase I)
Disease Control Rate (DCR) based on RECIST 1.1 criteria | 2 years
  DCR refers to Disease Control Rate. It is a measure used in clinical trials to indicate the proportion of patients whose cancer shrinks or remains stable over a specified period.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, China